CLINICAL TRIAL: NCT01582009
Title: A Phase I/II Study of the HDAC Inhibitor LBH-589 in Combination With the mTOR Inhibitor Everolimus (RAD001) in Metastatic Renal Cell Carcinoma
Brief Title: Panobinostat and Everolimus in Treating Patients With Metastatic or Unresectable Renal Cell Cancer That Does Not Respond to Treatment With Sunitinib Malate or Sorafenib Tosylate
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: pts off study, PI left institute
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I146308; NCI-2009-01599 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT01037257 (obsolete NCT alias)
Record Dates: First submitted 2010-07-15; First posted 2012-04-20 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Panobinostat; Everolimus; Chromatography, Liquid; Mass Spectrometry; Enzyme-Linked Immunosorbent Assay; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I: Oral Panobinostat and Oral Everolimus (Experimental): Patients receive oral panobinostat once daily on days 1, 3, 4, 8, 10, and 12 and oral everolimus once daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: panobinostat; Drug: everolimus; Other: laboratory biomarker analysis; Other: pharmacological study; Other: liquid chromatography; Other: mass spectrometry; Other: enzyme-linked immunosorbent assay; Other: immunohistochemistry staining method

INTERVENTIONS:
Drug: panobinostat — Given orally
  Other Names: Faridak; HDAC inhibitor LBH589; histone deacetylase inhibitor LBH589; LBH589
Drug: everolimus — Given orally
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: liquid chromatography — Correlative studies
  Other Names: LC
Other: mass spectrometry — Correlative studies
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry

SUMMARY:
RATIONALE: Panobinostat and everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving panobinostat together with everolimus and to see how well they work in treating patients with metastatic or unresectable renal cell cancer that does not respond to treatment with sunitinib malate or sorafenib tosylate

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability and determine the recommended dosing for the combination of LBH589 and Everolimus in patients with metastatic renal cell carcinoma. (Phase I) II. To assess the preliminary evidence of tumor response in patients treated with LBH589 and Everolimus. (Phase I) III. To evaluate the effect of LBH589 and Everolimus on the progression-free survival event rate. (Phase II) IV. To determine the clinical response rate of LBH589 and Everolimus in patients with metastatic renal cell carcinoma. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the toxicity of the combination of LBH589 and Everolimus in patients with metastatic renal cell carcinoma. (Phase II) II. To evaluate the effect of LBH589 and Everolimus on time-to-tumor-progression (TTP), disease-free survival and overall survival. (Phase II) III. To assess the pharmacodynamic effects of LBH589 and Everolimus in peripheral blood mononuclear cells (PBMNC) and tumor that are accessible before and after treatment, if available. (Phase II) IV. To evaluate the modulation of tumor metabolism and blood in patients treated with LBH589 and Everolimus by FDG and 015 water PET/CT scan. (Phase II)

OUTLINE: This is a dose-escalation study of panobinostat and everolimus, followed by a phase II study.

Patients receive oral panobinostat once daily on days 1, 3, 4, 8, 10, and 12 and oral everolimus once daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed metastatic or unresectable renal cell carcinoma
* Predominant clear cell component is required
* Patients must have metastatic disease which has progressed on or within 6 months of stopping treatment with VEGFR receptor tyrosine kinase inhibitors
* Previous therapy with bevacizumab, interleukin 2, or interferon alpha is also permitted
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Serum albumin >= 3g/dL
* AST/SGOT and ALT/SGPT =< 2.5 x upper limit of normal (ULN)
* Serum bilirubin =< 1.5 x ULN
* Serum creatinine =< 1.5 x ULN or 24-hour creatinine clearance >= 50 ml/min
* Serum potassium >= LLN
* Serum phosphorous >= LLN
* Serum total calcium (corrected for serum albumin) or serum ionized calcium >= LLN
* Serum magnesium >= LLN
* TSH and free T4 within normal limits (WNL); patients may be on thyroid hormone replacement
* ANC >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hb > 9 g/dL
* INR < 1.3 (or < 3 on anticoagulants)
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND fasting triglycerides =< 2.5 x ULN (in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Baseline MUGA or ECHO must demonstrate LVEF >= the lower limit of the institutional normal
* ECOG Performance Status of =< 2

Exclusion Criteria:

* Pure papillary and chromophobe renal cell carcinoma, collecting duct tumors and transitional cell carcinoma are not eligible
* Prior treatment with a pan-HDAC or mTOR inhibitor
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Patients who have had a major surgery of significant traumatic injury within 4 weeks of start of study drug and who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent; topical or inhaled corticosteroids are allowed
* Patients should not receive immunization with attenuated live vaccines within one weeks of study entry or during study period; close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus (Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY2a typhoid vaccines)
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* 1) Symptomatic congestive heart failure of New York Heart Association Class III or 4
* 2) Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* 3) Concomitant use of drugs with a risk of causing torsades de pointes
* 4) Severely impaired lung functions as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
* 5) Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN; optimal glycemic control should be achieved before starting trial therapy
* 6) Active (acute or chronic) or uncontrolled severe infections
* 7) Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis; a detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients; HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection
* A known HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods; adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug by both sexes
* Adults of reproductive potential who are not using effective birth control methods; if barrier contraceptive are being used, these must be continued throughout this trial by both sexes; hormonal contraceptives are not acceptable as a sole method of contraception
* Women of childbearing potential must have a negative urine or serum pregnancy test within 14 days prior to administration of everolimus
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus)
* Patients with a known hypersensitivity to everolimus (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients unwilling to or unable to comply with the protocol
* Patients currently receiving strong or moderate CYP3A4 inhibitors or inducers; patients should not begin study drugs until at least 72 hours after the last dose (or longer, as indicated) of the inhibitor or inducer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-03; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saby George, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Derived] Wood A, George S, Adra N, Chintala S, Damayanti N, Pili R. Phase I study of the mTOR inhibitor everolimus in combination with the histone deacetylase inhibitor panobinostat in patients with advanced clear cell renal cell carcinoma. Invest New Drugs. 2020 Aug;38(4):1108-1116. doi: 10.1007/s10637-019-00864-7. Epub 2019 Oct 25. PMID 31654285

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I: Oral Panobinostat and Oral Everolimus
Started | 26
Completed | 24
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Arm I: Oral Panobinostat and Oral Everolimus
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: 6 month PFS survival rate. Calculated as the total number of failures (deaths or progression) divided by the total follow-up or exposure time of patients on study. Assessed using Kaplan Meier and Proportional Hazards.
Time Frame: The time from registration to documentation of disease progression up to 3 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Oral Panobinostat and Oral Everolimus
Number analyzed (Participants) | 26
percentage of participants | 28 [11 to 48]

2. Primary Outcome: Number of Participants With Clinical Response
Description: Number of participants with clinical response. Response will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors ver 1.0 Committee [JNCI 92(3):205-216, 2000]. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST ver. 1.0 criteria.
Time Frame: The time from registration up to 3 years
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Oral Panobinostat and Oral Everolimus
Number analyzed (Participants) | 26
Participants | 0

3. Secondary Outcome: Number of Participants With an Adverse Event.
Description: Number of participants with an adverse event. Please refer to the adverse event reporting for more detail.
Time Frame: The time from registration up to 3 years
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Oral Panobinostat and Oral Everolimus
Number analyzed (Participants) | 26
Participants | 26

4. Secondary Outcome: Median Progression Free Survival
Description: Median progression free survival. Assessed using Kaplan Meier and Proportional Hazards.
Time Frame: The time from registration up to 3 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Oral Panobinostat and Oral Everolimus
Number analyzed (Participants) | 26
months | 5.3 [2.1 to 6.0]

5. Secondary Outcome: 6-month Overall Survival Rate
Description: 6-month overall survival rate
Time Frame: The time from registration up to 3 years
Population: All treated and eligible patients. Assessed using Kaplan Meier and Proportional Hazards.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Oral Panobinostat and Oral Everolimus
Number analyzed (Participants) | 26
percentage of participants | 96 [76 to 99]

ADVERSE EVENTS:
Arm/Group | Arm I: Oral Panobinostat and Oral Everolimus
Serious Adverse Events (participants affected / at risk) | 9/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Oral Panobinostat and Oral Everolimus (N=26)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (2)
Disease progression (General disorders) | 1 (2)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Confusional state (Psychiatric disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Oral Panobinostat and Oral Everolimus (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 (6)
Leukopenia (Blood and lymphatic system disorders) | 2 (4)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (28)
Atrial fibrillation (Cardiac disorders) | 2 (6)
Ocular hyperaemia (Eye disorders) | 1 (2)
Photophobia (Eye disorders) | 1 (2)
Visual impairment (Eye disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (8)
Abdominal pain lower (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 7 (22)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (4)
Flatulence (Gastrointestinal disorders) | 1 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 6 (16)
Stomatitis (Gastrointestinal disorders) | 3 (6)
Tongue ulceration (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (6)
Chills (General disorders) | 4 (8)
Fatigue (General disorders) | 14 (30)
Mucosal inflammation (General disorders) | 8 (20)
Oedema (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 5 (10)
Pain (General disorders) | 3 (8)
Pyrexia (General disorders) | 1 (2)
Cellulitis (Infections and infestations) | 1 (2)
Cystitis (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 1 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (2)
Urethritis (Infections and infestations) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 3 (8)
Blood albumin decreased (Investigations) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (6)
Blood calcium decreased (Investigations) | 1 (2)
Blood creatinine increased (Investigations) | 5 (16)
Blood fibrinogen increased (Investigations) | 1 (4)
Blood magnesium increased (Investigations) | 2 (4)
Blood phosphorus (Investigations) | 2 (6)
Blood phosphorus decreased (Investigations) | 2 (6)
Blood triglycerides increased (Investigations) | 5 (34)
Body temperature increased (Investigations) | 1 (2)
Electrocardiogram QT interval (Investigations) | 1 (2)
Electrocardiogram QT prolonged (Investigations) | 2 (4)
Gamma-glutamyltransferase increased (Investigations) | 2 (4)
Haemoglobin decreased (Investigations) | 4 (20)
High density lipoprotein decreased (Investigations) | 1 (2)
Low density lipoprotein increased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (2)
Protein total increased (Investigations) | 1 (2)
White blood cell count decreased (Investigations) | 1 (12)
Decreased appetite (Metabolism and nutrition disorders) | 4 (10)
Dehydration (Metabolism and nutrition disorders) | 1 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (12)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (26)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (12)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Dysgeusia (Nervous system disorders) | 2 (4)
Headache (Nervous system disorders) | 4 (10)
Hemicephalalgia (Nervous system disorders) | 1 (2)
Hypogeusia (Nervous system disorders) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 3 (6)
Insomnia (Psychiatric disorders) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (2)
Nocturia (Renal and urinary disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (8)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (6)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (2)
Embolism (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 3 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes